CLINICAL TRIAL: NCT03355625
Title: Platelet Function During Extracorporeal Membrane Oxygenation in Adult Patients
Status: Completed | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Collaborators: University of Aarhus (Other)
Responsible Party: Sponsor
Organization: University of Aarhus (Other)
Other Study IDs: ECMO-Camilla
Record Dates: First submitted 2017-11-22; First posted 2017-11-28 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Extracorporeal Membrane Oxygenation; Platelet Activation; Platelet Aggregation; Platelet Function Tests; Blood Platelets; Intensive Care Units
Keywords: Flow Cytometry; eCPR; Extracorporeal Life Support

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary aim is to describe platelet function in adult patients treated with extracorporeal membrane oxygenation (ECMO). A clarification of the platelet function in these critically ill patients contributes to an understanding of the mechanisms underlying their coagulopathy.

The present study is a substudy to the study entitled; "Coagulopathy During Extracorporeal Membrane Oxygenation" (pending Clinical Trial ID number).

DETAILED DESCRIPTION:
The knowledge of platelet function during extracorporeal membrane oxygenation (ECMO) remains sparse. In the present study, the aim is to investigate platelet function in adult patients treated with ECMO using flow cytometry. The investigators hypothesize that platelet function increases from day 1 to day 3 in patients treated with ECMO. The secondary aim is to investigate the association between platelet function and the incidence of bleeding episodes and thrombosis during ECMO treatment.

The present study is a substudy to the study entitled; "Coagulopathy During Extracorporeal Membrane Oxygenation" (pending Clinical Trial ID number).

ELIGIBILITY:
Inclusion Criteria:

* Treatment with veno-venous or veno-arterial ECMO
* Age ≥18 years

Exclusion Criteria:

* ECMO treatment initiated post-operatively

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with ECMO at the Intensive Care Unit East, Aarhus University Hospital.
Sampling Method: Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Changes in platelet function | Platelet function measured day 1 and day 3 on ECMO
  Platelet function on day 3 compared with day 1 on ECMO. Measured by flow cytometry

SECONDARY OUTCOMES:
Changes in platelet aggregation | Platelet function measured every morning from day 1 to day 8 on ECMO (except weekends).
  Comparison of platelet aggregation measured by whole blood impedance aggregometry (Multiplate).
Immature platelet count | Measured every morning from day 1 to day 8 on ECMO (except weekends)
  Estimation of platelet turn-over measured by a blood analyzer (Sysmex)
Platelet count | Measured every morning from day 1 to day 8 on ECMO (except weekends)
  Estimation of platelet count measured by a blood analyzer (Sysmex)

CONTACTS AND LOCATIONS:
Overall Officials: Camilla Mains Balle, Research fellow, Principal Investigator — Centre of Haemophilia and Thrombosis, Department of Clinical Biochemistry, Aarhus University Hospital; Anne-Mette Hvas, Professor, MD, PhD, Study Chair — Centre of Haemophilia and Thrombosis, Department of Clinical Biochemistry, Aarhus University Hospital; Anni Nørgaard Jeppesen, MD, PhD, Study Chair — Department of Anaesthesiology and Intensive Care Unit East, Aarhus University Hospital; Steffen Christensen, MD, PhD, Study Chair — Department of Anaesthesiology and Intensive Care Unit East, Aarhus University Hospital
Locations (2):
- Denmark (2):
  - Centre of Haemophilia and Thrombosis, Department of Clinical Biochemistry, Aarhus University Hospital, Aarhus
  - Department of Anaesthesiology and Intensive Care Unit East, Aarhus University Hospital, Aarhus

IPD SHARING:
Plan to Share IPD: No